CLINICAL TRIAL: NCT06244979
Title: iMagIng pulmonaRy Aspergillosis Using Gallium-68-dEferoxamine
Acronym: MIRAGE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 115136; 2023-509744-10-00 (Other: CTIS nr)
Record Dates: First submitted 2024-01-03; First posted 2024-02-06 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Aspergillosis; Chronic Pulmonary Aspergillosis; Allergic Bronchopulmonary Aspergillosis
MeSH Terms: conditions — Pulmonary Aspergillosis; Aspergillosis, Allergic Bronchopulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Patients will undergo a PET/CT scan at t=60 min after a single intravenous injection of a fixed dose of 100 MBq +/- 10% [68Ga]Ga-DFO-B (gallium-68-deferoxamine) which contains 100 µg deferoxamine (DFO-B).
  Interventions: Other: Radiopharmaceutical: gallium-68-deferoxamine ([68Ga]Ga-DFO-B)

INTERVENTIONS:
Other: Radiopharmaceutical: gallium-68-deferoxamine ([68Ga]Ga-DFO-B) — 100 MBq +/- 10% [68Ga]Ga-DFO-B which contains 100 µg DFO-B (see description in arm description)

SUMMARY:
This is a single center open-label feasibility trial involving a single study visit for participants. The purpose of the study is to demonstrate the feasibility of [68Ga]Ga-DFO-B PET/CT (gallium-68-deferoxamine) for the visualization of pulmonary Aspergillus infection.

The incidence of fungal infections is on the rise and are associated with significant mortality. Diagnosis pulmonary aspergillosis can be can be challenging, often requiring invasive tests such as bronchoscopy and lung tissue biopsies. Molecular imaging, specifically using radiolabeled siderophores like [68Ga]Ga-DFO-B, offers a non-invasive and location-specific approach to visualize and evaluate infections. Siderophores, critical for pathogenic microbes like Aspergillus fumigatus, play a role in iron acquisition. Preclinical studies with radiolabeled deferoxamine (DFO-B) demonstrated distinct accumulation at infection sites. Additionally, [68Ga]Ga-DFO-B PET/CT may differentiate between Aspergillus infection and cancer, making it a promising non-invasive diagnostic tool for pulmonary aspergillosis.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is at least 18 years old on the day of inclusion.
2. The patient has suspected chronic pulmonary aspergillosis or ABPA.
3. There is no significant interference with standard care and follow-up.

Exclusion Criteria:

1. The patient is pregnant or planning on becoming pregnant.
2. The patient has severe kidney dysfunction with eGFR < 30 ml/min/kg and/or receives dialysis.
3. The patient has (chronic) iron overload.
4. The patient has been receiving antifungal treatment for more than 48 hours prior to the study day.
5. The patient is not able to lie still in the scanner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake values (SUV) of [68Ga]Ga-DFO-B | PET/CT will be performed 60 minutes after intravenous injection of [68Ga]Ga-DFO-B
  Measurement of the amount of radiotracer uptake ([68Ga]Ga-DFO-B) in suspected Aspergillus lesions in patients with pulmonary aspergillosis.
Target-to-background ratios of [68Ga]Ga-DFO-B | PET/CT will be performed 60 minutes after intravenous injection of [68Ga]Ga-DFO-B
  Ratio of the signal intensity or uptake in suspected Aspergillus lesions (target) to the background signal intensity in the surrounding normal tissues in patients with pulmonary aspergillosis.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Brüggemann, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- RadboudUMC, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No